CLINICAL TRIAL: NCT00731276
Title: Phase I Study to Investigate Genotype-based Dose Individualization of Irinotecan in Asian Cancer Patients
Brief Title: Irinotecan in Treating Asian Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000601207; SINGAPORE-NCC0703
Record Dates: First submitted 2008-08-07; First posted 2008-08-08 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Irinotecan; Pharmacogenomic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Four Regimens (Other): The study has four type of regimens, and dosing of irinotecan depends on genotype of patient.
  Four Regimens are:
  1. Weekly Irinotecan (Irinotecan given at day 1, 8 and 15) every four weekly
  2. Weekly Xeliri ( Irinotecan given at day 1, 8 and 15)+ (Xeloda tabs 2000mg/m2 consumed over 14 days) every three weekly
  3. Three-weekly Xeliri (Irinotecan given at day 1 only) + (Xeloda tabs 2000mg/m2 consumed over 14 days) every three weekly
  4. Two-weekly FOLFIRI (Irinotecan given at day 1 only) + (CI Fluorouracil 600mg/m2 over 22hrs, IV Folinic Acid 200mg/m2 over 2hrs and IVP Fluorouracil 400mg/m2) every two weekly
  Interventions: Drug: irinotecan hydrochloride; Other: pharmacogenomic studies; Other: pharmacological study

INTERVENTIONS:
Drug: irinotecan hydrochloride
Other: pharmacogenomic studies
Other: pharmacological study

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase I trial is studying the side effects and best dose of irinotecan in treating Asian patients with solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the dose-limiting toxicity and maximum tolerated dose of irinotecan hydrochloride according to the genotype status of Asian patients with solid tumors.

Secondary

* To investigate the pharmacokinetics of irinotecan hydrochloride and its metabolites SN-38 and SN-38G.
* To evaluate time to tumor response, response duration, and time to progression in these patients.

OUTLINE: Patients are stratified according to genotype status (UGT1A1*28 vs UGT1A1*6)

Patients receive irinotecan hydrochloride IV once weekly for 3 weeks. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo blood sample collection periodically for pharmacogenetic, pharmacokinetic, and pharmacodynamic studies.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed solid tumors

  * Failed at least one line of prior chemotherapy
* Must belong to either Chinese, Malay, or Indian ethnic groups
* Previously irradiated disease allowed provided marker lesions not within the irradiated field
* Presence of at least one bidimensionally measurable, non-CNS indicator lesion, defined by radiologic study (including CT or MRI scan, ultrasound, or chest X-ray) or physical exam, meeting 1 of the following criteria:

  * Measurable disease on CT or MRI scan must have one diameter ≥ 1 cm and one diameter ≥ 2 cm
  * Measurable disease on chest X-ray or ultrasound must have both diameters ≥ 2 cm
  * Palpable tumor masses that cannot be evaluated radiologically must have two diameters ≥ 2 cm
  * Measurable skin lesion must have at least one diameter ≥ 1 cm
* No unidimensionally measurable or evaluable only disease
* No known brain or leptomeningeal metastasis
* No uncontrolled large pleural effusions

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 3 months
* Absolute granulocyte count ≥ 1,000/µL
* WBC ≥ 3,500/µL
* Hemoglobin ≥ 9 g/dL
* Platelet count ≥ 100,000/µL
* Serum total bilirubin ≤ 2.0 mg/dL
* ALT/AST < 2.5 times normal (5 times normal in patients with known metastatic disease in the liver)
* Creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No medical problems severe enough to prevent compliance with the study requirements
* No prior malignancies, except for adequately treated basal cell or squamous cell carcinoma, carcinoma in situ of the cervix, or other cancer for which the patient has been disease-free for 5 years
* No active or uncontrolled infection
* No pre-existing cardiac disease, including congestive heart failure, arrhythmia requiring treatment, or myocardial infarction within the past 3 months
* No pneumonitis
* No uncontrolled diabetes mellitus (i.e., random blood glucose > 200 mg/dL)
* No inflammatory bowel disease

PRIOR CONCURRENT THERAPY:

* At least 1 week since prior and no concurrent ketoconazole
* More than 4 weeks since prior chemotherapy or radiotherapy
* At least 2 weeks since prior and no concurrent Hypericum perforatum (St. John wort)
* No prior irinotecan hydrochloride
* No concurrent investigational antineoplastic therapy or other investigational drugs

Ages: 21 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-04-03 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity | No time frame defined. Trial is still recruiting.
Maximum tolerated dose | No time frame defined. Trial is still recruiting.

SECONDARY OUTCOMES:
Pharmacokinetics | No time frame defined. Trial is still recruiting.
Time to tumor response | No time frame defined. Trial is still recruiting.
Time to progression | No time frame defined. Trial is still recruiting.
Response duration | No time frame defined. Trial is still recruiting.

CONTACTS AND LOCATIONS:
Overall Officials: Su Pin Choo, MD, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre - Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No